CLINICAL TRIAL: NCT00133354
Title: Double-blind Trial Investigating the Safety and Efficacy of the Inhibitor Anastrozole (ARIMIDEX) in Delaying Epiphyseal Fusion and Increasing Height Potential of Adolescent Males With Growth Hormone (GH) Deficiency
Brief Title: Arimidex Multicenter Trial in Growth Hormone (GH) Deficient Boys
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: AstraZeneca (Industry); Genentech, Inc. (Industry); EMD Serono (Industry)
Responsible Party: Principal Investigator, Nelly Mauras, Chief, Division of Endocrinology, Diabetes & Metabolism, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: IRUSANAS0008; M2372s; 23381
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Hypopituitarism
Keywords: Puberty; Growth hormone deficiency; aromatase inhibitors; estrogen; bone mineral density; short stature
MeSH Terms: conditions — Hypopituitarism; Dwarfism, Pituitary; Dwarfism | interventions — Anastrozole; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arimidex and Growth Hormone (Active Comparator)
  Interventions: Drug: Arimidex (Anastrozole); Drug: Growth Hormone
- Placebo and Growth Hormone (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Growth Hormone

INTERVENTIONS:
Drug: Arimidex (Anastrozole) — Subjects will be randomized in a 1:1 ratio to be given either Arimidex 1 mg or placebo orally. Subjects will receive trial treatment for 36 months while continued on GH.
  Arms: Arimidex and Growth Hormone
Drug: Placebo — Subjects will be randomized in a 1:1 ratio to be given either Arimidex 1 mg or placebo orally. Subjects will receive trial treatment for 36 months while continued on GH.
  Arms: Placebo and Growth Hormone
Drug: Growth Hormone — GH (Nutropin®, Genentech, So. San Francisco, CA) will be administered throughout the trial at a dose of ~0.3mg/kg.w (no more than 0.4mg/kg.w) given subcutaneously (SC) at bedtime daily. Dose adjustments on the GH dose will be made by the investigator at least every 6mo.

SUMMARY:
The purpose of this study is to see if Arimidex, an aromatase inhibitor, can delay epiphyseal fusion and increase predicted adult height in boys who are growth hormone deficient, in puberty, and who are taking growth hormone. This is a double blind, placebo controlled 3 year trial.

ELIGIBILITY:
Inclusion Criteria:

* Growth hormone deficient by formal testing with two provocative agents.
* Treated with growth hormone for a minimum of 6 months prior to study entry.
* Growth hormone doses must be maintained at 0.2-0.4mg/kg/wk while in protocol.
* Stable organic pathology
* Presence of puberty [genital Tanner Stage > II (>4cc testicular volume)]
* Bone age (BA) > or = 11.5 years and < 15 years

Exclusion Criteria:

* Participation in any other trial involving hormone therapy for at least 6 months prior.
* Chronic illnesses requiring long term medication that impair growth. (Stable patients with occasional asthma, patients on Ritalin or Adderall or patients on topical acne medication may be included).
* Hereditary disease diagnosed clinically.
* Moderate to severe scoliosis.

Ages: 11 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2001-11; Primary Completion 2006-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The primary measure of efficacy is change in predicted adult height based on rate of bone age advancement. | 12months, 24months, 36months

SECONDARY OUTCOMES:
The secondary objective is to determine the effect of Arimidex® treatment in bone mineralization in pubertal GH deficient males treated concurrently with growth hormone. | 12months, 24months, 36months

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States